CLINICAL TRIAL: NCT05648734
Title: Impact of Anti-Inflammatory and Anti-Fibrotic Drugs on Post-acute COVID-19 Pulmonary Fibrosis
Brief Title: Anti-Inflammatory and Anti-Fibrotic Drugs in Post COVID-19 Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MD.21.09.526 - 2021/09/12
Record Dates: First submitted 2022-11-30; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Post-COVID-19 Syndrome; Lung Fibrosis
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Pulmonary Fibrosis | interventions — Adrenal Cortex Hormones; Colchicine; pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: Patients received Corticosteroids only
  Interventions: Drug: Corticosteroids alone
- Group B: Patients received Corticosteroids in combination with Colchicine
  Interventions: Drug: Corticosteroids + Colchicine
- Group C: Patients received Corticosteroids in combination with Pirfenidone
  Interventions: Drug: Corticosteroids + Pirfenidone
- Group D: Patients received Corticosteroids in combination with Colchicine and Pirfenidone
  Interventions: Drug: Corticosteroids + Colchicine + Pirfenidone for ≥ 14 days

INTERVENTIONS:
Drug: Corticosteroids alone — (≥ 20 mg prednisolone or its equivalent for ≥ 10 days after hospital discharge)
  Other Names: Solupred; Disperlone; Methabiogen; Epicopred
  Groups: Group A
Drug: Corticosteroids + Colchicine — (≥ 20 mg prednisolone or its equivalent for ≥ 10 days) + Colchicine (1 mg/day for ≥ 10 days)
  Groups: Group B
Drug: Corticosteroids + Pirfenidone — (≥ 20 mg prednisolone or its equivalent for ≥ 10 days) + Pirfenidone (267 mg TID for ≥ 14 days)
  Other Names: Corticosteroids + Pirfinix
  Groups: Group C
Drug: Corticosteroids + Colchicine + Pirfenidone for ≥ 14 days — (≥ 20 mg prednisolone or its equivalent for ≥ 10 days) + Colchicine (1 mg/day for ≥ 10 days) + Pirfenidone (267 mg TID for ≥ 14 days)
  Groups: Group D

SUMMARY:
In this study we aim to evaluate the radiological and functional changes in post-acute covid-19 pulmonary fibrosis patients in relation to anti-inflammatory and/or antifibrotic drugs prescribed during and after covid-19 pneumonia.

DETAILED DESCRIPTION:
This study is a prospective and retrospective cohort study in which post COVID-19 patients who are following up at post COVID-19 clinic are evaluated regarding presence and degree of Post COVID-19 Pulmonary Fibrosis (PCPF) in relation to anti-inflammatory and/or anti-fibrotic drugs.

Adult patients who have COVID-19 pneumonia confirmed either by RT-PCR or radiologically by CT scan and according to WHO severity classification are (Moderate, severe, or critical) and has received either:

* Corticosteroids alone (≥ 20 mg prednisolone or its equivalent for ≥ 10 days after hospital discharge) - Group A.
* Corticosteroids in combination with Colchicine (1 mg/day for ≥ 10 days) - Group B.
* Corticosteroids in combination with Pirfenidone (267 mg TID for ≥ 14 days) - Group C.
* Corticosteroids in combination with Colchicine and Pirfenidone (for ≥ 14 days) - Group D.

Pulmonary function test: Spirometry: measurement of lung volumes and capacities (forced expiratory volume in first second FEV1, Forced Vital Capacity FVC, FEV1/FVC and FEF25/75) after 1 month and 3 months of the onset of symptoms.

Radiological scoring: Baseline High resolution CT scan of the chest will be performed at baseline, 1 month and 3 months after onset of symptoms. Chest CT-Severity Scoring (Chest CT-SS) for assessing COVID-19 burden on the initial scan will be calculated. This score uses lung opacification as a surrogate for extension of the disease in the lungs. According to the anatomic structure, the 18 segments of both lungs were divided into 20 regions, in which the posterior apical segment of the left upper lobe was subdivided into apical and posterior segmental regions, whereas the anteromedial basal segment of the left lower lobe was subdivided into anterior and basal segmental regions. The lung opacities in all the 20 lung regions were subjectively evaluated on chest CT images using a system attributing score of 0, 1, and 2 if parenchymal opacification involved 0%, less than 50%, or equal to or more than 50% of each region, respectively. The CT-SS was defined as the sum of the individual scores in the 20 lung segment regions, which may range from 0 to 40 points

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have COVID-19 pneumonia confirmed either by RT-PCR or radiologically by CT scan and according to WHO severity classification are (Moderate, severe, or critical) and has received either: Corticosteroids alone.
* Corticosteroids in combination with Colchicine.
* Corticosteroids in combination with Pirfenidone.
* Corticosteroids in combination with Colchicine and Pirfenidone.

Exclusion Criteria:

* None COVID-19 pneumonia.
* Patients with previous parenchymal lung disease.
* Patients receiving anti-fibrotic or anti-inflammatory drugs due to other chronic disease.
* Patients who received anti-fibrotic and or ant inflammatory drugs for duration and or doses less than presumed or those who reported noncompliance to treatment.
* Patients with uncontrolled comorbidities.
* Patients who develop severe intolerable side effects or derangement of liver enzymes more than 5 folds.
* Pregnant ladies with COVID-19 pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort study in which post COVID-19 patients who are following up at post COVID-19 clinic are evaluated regarding presence and degree of Post COVID-19 Pulmonary Fibrosis (PCPF) in relation to anti-inflammatory and/or anti-fibrotic drugs.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary Functions Test | 8 weeks
  Change in FVC from 1 month to 3 months follow up after hospital discharge
Radiological scoring | 8 weeks
  Change in Chest CT Severity Scoring (Chest CT-SS) from 1 month to 3 months follow up after hospital discharge compared to baseline CT Chest scan

CONTACTS AND LOCATIONS:
Overall Officials: Amina Abdel Maksoud, MD, Study Director — Mansoura University, Faculty of Medicine; Dalia Fahmy, MD, Study Director — Mansoura University, Faculty of Medicine; Aida Yousef, MD, Study Director — Mansoura University, Faculty of Medicine; Mohamed Tohlob, MD, Study Director — Mansoura University, Faculty of Medicine
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Anonymous'd individual data will be available with the corresponding author on reasonable request